CLINICAL TRIAL: NCT04539613
Title: Controlled Ovarian Hyperstimulation (COH) With Sequential HPFSH & HMG Versus Rec-F.S.H Alone in ICSI Cycle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alaa Fouli Gaber Ebrahim (Other)
Responsible Party: Sponsor-Investigator, Alaa Fouli Gaber Ebrahim, Controlled Ovarian Hyperstimulation (COH) With Sequential HPFSH & HMG Versus Rec-F.S.H Alone in ICSI Cycle, Minia University
Organization: Minia University (Other)
Other Study IDs: COH in ICSI
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Stimulation in ICSI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group1: Group 1(50 case) which will receive hp FSH (fostimon ibsa) (150 IU per ampoule)will be started on day 2 of menstruation and then after six days, HMG (meriofert ibsa), 150 Iu, s.c) will be added
  Interventions: Drug: HPFSH & HMG
- group2: Group 2(50 case) will be treated with recombinant FSH alone (Gonal-F) (150 IU per ampoule)

INTERVENTIONS:
Drug: HPFSH & HMG — . Various gonadotropin preparations
  Other Names: rec-F.S.H
  Groups: group1

SUMMARY:
despite the large number of papers published on COH protocols comparing the efficiency of different exogenous gonadotropins, no confirmed protocol exists, and it is not quite clear which is superior to the others.

DETAILED DESCRIPTION:
, the objective of the current study was to compare the efficacy of 2 different ovarian stimulation protocols, comprising hpFSH, HMG versus R-FSH on oocyte and embryo quality and IVF treatment outcome in patients undergoing IVF or intracytoplasmic sperm injection (ICSI)(4).

ELIGIBILITY:
Inclusion Criteria:

* 1-Aged 20-35 yr, male factor, 2-Tubal or unexplained infertility, 3-regular menstruation cycle between 21 and 35 days, 4-Normal function of uterus according to hysterosalpingography, hysteroscopy or transvaginal ultrasonography, 5-Normal ovaries according to transvaginal ultrasonography during past 6 months prior to study and compatible with normal adnexa and 6-Normal ovarian anatomy, and serum FSH level less than 8 IU/l All women showed no recognizable endometriosis according to symptoms and clinical examination in transvaginal ultrasonography or diagnostic laparoscopy. 7-7-All women have a history of unexplained infertility 8-Normal ovulatory function and normal semen analysis according to the World Health Organization criteria .

Exclusion Criteria:

* Patients with other ovulation disorders such as hypo and hypergonadotropic, hypogonadism, hyperprolactinemia.

  2-Thyroid disorders. 3-Ovarian or adrenal neoplasms. 4-Cushing syndrome. 5-previous history of systemic diseases such as endocrine and metabolic disorders.

  6- Previous history of inappropriate ovarian response to stimulation with gonadotropins (poor responders).

  7-Prior history of more than 3 unsucce

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Normal ovulatory function and normal semen analysis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
fertility outcomes (pregnancy rate, abortion and live birth rate) in IVF patients. | 5months
  (pregnancy rate, abortion and live birth rate) in IVF patients.

CONTACTS AND LOCATIONS:
Locations (1):
- El neel, Minya, Egypt

REFERENCES:
- [Background] Kamel RM. The onset of human parturition. Arch Gynecol Obstet. 2010 Jun;281(6):975-82. doi: 10.1007/s00404-010-1365-9. Epub 2010 Feb 3. PMID 20127346